CLINICAL TRIAL: NCT04108572
Title: The Choosing Healthy Eating for Infant Health (CHErIsH) Study
Acronym: CHErIsH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: National University of Ireland, Galway, Ireland (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Patricia Kearney, Principle Investigator, University College Cork
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HRB_CHErIsH
Record Dates: First submitted 2019-05-24; First posted 2019-09-30 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Pediatric Obesity
Keywords: Child Obesity; Infant Feeding; Feasibility study
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Non-randomised feasibility study of an infant feeding intervention and implementation strategy, with embedded process evaluation and economic evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infant feeding intervention (Experimental): The intervention will be delivered to parents by practice nurses and/or GPs in MPHC at each of the vaccination visits, prior to administration of the vaccination. These vaccination visits take place at 2, 4, 6, 12 and 13 months. This intervention consists of 1) verbally delivered pre-specified infant feeding messages, and 2) provision of additional infant-feeding resources including an information leaflet, a magnet, an infant bib and access to an informational website.
  Interventions: Behavioral: Infant feeding

INTERVENTIONS:
Behavioral: Infant feeding — Verbally delivered pre-specified infant feeding message. The messages focus on appropriate milk feeding and establishing complementary feeding and solid food introduction in relation to timing and practical guidance around processes of feeding and provision of additional infant-feeding resources including information leaflet, a magnet, an infant bib and access to an informational website.

SUMMARY:
The Choosing Healthy Eating for Infant Health (CHErIsH) intervention is a complex infant feeding intervention delivered at infant vaccination visits, alongside a healthcare professional (HCP) level implementation strategy to support delivery. The primary aim of CHErIsH pilot feasibility study is to collect and examine data on the acceptability and feasibility of the delivery of the brief infant-feeding intervention by HCPs to parents at child vaccination visits, and the strategy to support the implementation of this intervention in primary care for HCPs. Furthermore, half of all potential participants will be invited to provide maternal and infant biomarkers and/or take part in SWAT (study within a trial) which includes questions about infant feeding that were put together as part of a Core Outcome Set. These questions are important as they give a better understanding about what works and what doesn't. This will facilitate the refinement of the intervention and its implementation strategy, and inform the next step of the CHErIsH study, such as a definitive trial.

DETAILED DESCRIPTION:
The Choosing Healthy Eating for Infant Health (CHErIsH) intervention is a non-randomised feasibility study of an infant feeding intervention and implementation strategy, with embedded process evaluation and economic evaluation.

The CHErIsH feasibility study will address the following research questions:

1. Are the intervention content, delivery and implementation procedures acceptable to parents who will receive the intervention, and HCPs who will deliver the intervention?
2. Are the data collection processes, including mode and duration of data collection and outcome measures used, acceptable to parents and HCPs?
3. Is the intervention feasible to deliver in primary care practice, in terms fidelity of delivery and receipt of the intervention?
4. Is the study feasible in terms of recruitment and retention procedures and data collection?
5. What are the costs associated with the intervention and its implementation strategy?

ELIGIBILITY:
Inclusion Criteria (Health care professionals):

* Involved in the delivery of routine infant vaccinations
* Completed training to deliver the intervention.

Inclusion Criteria (Parents):

* Parent of an infant ≤ 6 weeks of age at study recruitment.
* Intends to attend a participating GP and/or PN in the primary care centre for child's vaccination visits.
* Is over 18 years of age.
* Can provide written informed consent to participate.

Exclusion Criteria:

* n/a

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Parent intervention feedback | Tp3= at infant's 13 month vaccination visit.
  Four-item measures of implementation outcomes including Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), Feasibility of Intervention Measure (FIM) will be used together to assess the acceptability, appropriateness and feasibility of the parent-level intervention (following intervention cessation). Scale values range from 1 to 5. 1 = completely disagree and 5 completely agree.
Healthcare professional intervention feedback | Tp3= at infant's 13 month vaccination visit.
  Four-item measures of implementation outcomes including Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), Feasibility of Intervention Measure (FIM) will be used together to assess the acceptability, appropriateness and feasibility of the parent-level intervention (following intervention cessation). Scale values range from 1 to 5. 1 = completely disagree and 5 completely agree.

SECONDARY OUTCOMES:
Intervention reach and recruitment | Tp1= baseline, prior to infant's 2-month vaccination visit; Tp2= by the infant's 6-month vaccination visit); Tp3= at infant's 13 month vaccination visit.
  Number of invitations sent to parents, acceptances to participate, and refusals
Appropriateness of parent data collection processes and outcome measures | Tp1= baseline, prior to infant's 2-month vaccination visit; Tp2= by the infant's 6-month vaccination visit); Tp3= at infant's 13 month vaccination visit.
  Number of missing items self report questionnaires and follow-up rates
Parent intervention fidelity | Tp3= at infant's 13 month vaccination visit.
  Checklist assessing intervention components received by parent (e.g., 'Did you receive a leaflet about infant feeding?').
Healthcare professional intervention fidelity | Tp3= at infant's 13 month vaccination visit.
  Checklist assessing intervention components delivered by HCPs (e.g., 'Did you provide parent with a leaflet about infant feeding?').
Estimate of resources and costs needed to deliver the intervention | Tp3= at infant's 13 month vaccination visit.
  Resources in relation the intervention will be identified. Costs incurred as a consequence of the intervention and implementation strategy will be identified. This will include all time and resources expended, and costs borne by Healthcare Centre including the training and time spent by healthcare professionals and administrative staff involved in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Patricia Kearney, Principal Investigator — University College Cork
Locations (1):
- Mallow Primary Health Care Centre, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Queally M, Doherty E, Finucane FM, O'Neill C. Low expectations: Do teachers underestimate the ability of overweight children or the children of overweight mothers? Econ Hum Biol. 2017 Nov;27(Pt A):26-32. doi: 10.1016/j.ehb.2017.04.006. Epub 2017 Apr 28. PMID 28486211
- [Background] Black L, Matvienko-Sikar K, Kearney PM. The association between childcare arrangements and risk of overweight and obesity in childhood: a systematic review. Obes Rev. 2017 Oct;18(10):1170-1190. doi: 10.1111/obr.12575. Epub 2017 Jul 4. PMID 28677302